CLINICAL TRIAL: NCT04178005
Title: Cladribine Tablets After Treatment With Natalizumab (CLADRINA)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Olaf Stuve, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2019-1618
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cladribine (Other): All study participants will receive treatment with cladribine 10 mg tablets at the recommended cumulative dose of 3.5 mg/kg, divided into 2 yearly treatment courses (1.75 mg/kg per treatment course). This regimen corresponds to the recommended dosage as per the USPI.
  Each treatment course is divided into 2 treatment cycles:
  * Administration of first treatment course (year 1 treatment):
  * First cycle: Starts on Day 1 of the study
  * Second cycle: Administered 23 to 27 days after the last dose of first cycle.
  * Administration of second treatment course (year 2 treatment):
  * First cycle: Administered at least 43 weeks after the last dose of year 1 treatment
  * Second cycle: Administered 23 to 27 days after the last dose of first cycle of year 2 treatment.
  The cycle dosage will be administered as 1 or 2 cladribine 10 mg tablets daily over 4 or 5 consecutive days.
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — All study participants will receive treatment with cladribine 10 mg tablets at the recommended cumulative dose of 3.5 mg/kg, divided into 2 yearly treatment courses (1.75 mg/kg per treatment course). This regimen corresponds to the recommended dosage as per the USPI
  Other Names: Mavenclad

SUMMARY:
The purpose of this study is to generate hypotheses regarding the safety, efficacy, and immunological impact of cladribine tablets after treatment with natalizumab in patients with relapsing-remitting multiple sclerosis (RRMS) and active secondary progressive multiple sclerosis (active SPMS).

DETAILED DESCRIPTION:
This will be an open label, single arm, multicenter, collaborative phase 4 research study, designed to generate hypotheses regarding the transition to cladribine tablets after treatment with natalizumab in patients with relapsing forms of multiple sclerosis MS, to include relapsing-remitting multiple sclerosis (RRMS) and active secondary progressive multiple sclerosis (SPMS).

The total duration of this interventional study will be 2 years, but patients who require additional time (up to 6 months) for recovery of Absolute lymphocyte count (ALC) to 800 cells/ul prior to the second treatment course will be followed for up to 6 additional months in order to have a full second year of follow up after initiation of the second year's treatment course (for a total study duration of up to 30 months in some patients). A total of 40 study participants with relapsing forms of MS, to include RRMS and active SPMS, who meet the criteria for treatment with cladribine tablets as per the approved United States Prescribing Information (USPI) are planned to be enrolled at up to three centers in the United States. All study participants will receive treatment with cladribine 10 mg tablets during year 1 and year 2 according to the approved USPI (EMD Serono, 2019). Cladribine 10 mg tablets will be provided as commercial material. Treatment with cladribine tablets is intended to be initiated approximately 14 days after the last infusion of natalizumab (e.g., a 14-day "washout"), with a maximum permissible washout period of no more than four weeks.

After successful completion of the study, all participants in CLADRINA will be offered to participate in the CLADRINA 2-Year Extension study. During this extension trial, there will be no intervention. Patient will be followed for an additional 24 months, and their clinical and paraclinical disease activity will be assessed through neurological examinations, EDSS scores, brain MRI, and biological markers.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following inclusion criteria will be eligible for enrollment in the study:

1. Age between 18 and 60 years, inclusive.
2. Diagnosis of relapsing forms of MS, to include RRMS and active SPMS, diagnosed with McDonald Criteria 2005, 2010, and/or 2017 (1-3)
3. EDSS 0 - 5.5 (Functional system changes in cerebral (or mental) functions and in bowel and bladder functions not used in determining EDSS for protocol eligibility).
4. Has had a minimum of 12 months of continuous natalizumab therapy (300 mg/d), including patients receiving extended interval dosing of natalizumab (e.g., less frequently than every-4-week infusion).
5. Negative history for any relapses at least 28 days prior to enrollment.
6. Weighing between 40 kilograms or more.
7. Female subjects of childbearing potential must use effective methods of contraception to prevent pregnancy for 4 weeks before initiation of cladribine tablets and must agree to continue to practice adequate contraception for at least 6 months after the last dose. Women using systemically acting hormonal contraceptives should add a barrier method during cladribine treatment and for at least 4 weeks after the last dose in each treatment year.
8. Female subjects must not be pregnant; female subjects must not be lactating or breast-feeding at least 10 days after the last dose.
9. Male subjects must be willing to use a condom during dosing and for six months after the last dose. Alternatively, their female partner must use another form of contraception (such as an intra-uterine device [IUD], barrier method with spermicide, or hormonal contraceptive [e.g., implant, injectable, patch or oral]) during dosing and for six months after last dose.
10. Understands and is capable of following through with study protocol requirements and assessments.
11. Willing to provide voluntary and informed consent based on the Health Insurance Portability and Accountability Act (HIPPA).

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will not be eligible for enrollment in the study:

1. Natalizumab failure based on clinician's discretion.
2. Not active progressive MS (4).
3. A diagnosis of PML or any suspicion of PML.
4. A diagnosis of Clinically Isolated Syndrome
5. Known hypersensitivity to cladribine.
6. Any prior exposure to cladribine.
7. Lymphocyte count not within normal limits of the local, hospital laboratory.
8. Previous or current exposure to mitoxantrone, azathioprine, methotrexate, cyclophosphamide, myelosuppressive treatments, total lymphoid irradiation.
9. Receiving oral or systemic corticosteroid treatments within the 28 days prior to enrollment.
10. Receiving cytokine base treatment, Intra Venous Immuno Globulin (IVIG) or Plasma pheresis, 3 months prior to enrollment in the study.
11. Having platelet count or neutrophil count below the lower limit of the normal range within the 28 days prior to enrollment in the study.
12. Positive for HIV, or positive hepatitis C antibody test or hepatitis B surface antigen test and/or core antibody test for IgG and/or IgM.
13. History of tuberculosis (TB), presence of active tuberculosis, or latent tuberculosis as detected by local standard of practice like imaging (e.g., chest X-ray, chest CT scan, MRI) and/or positive QuantiFERON-TB Gold test and/or skin test and/or clinical examination or has had latent TB disease at any time in the past.
14. Immunocompromised subjects, including subjects currently receiving immunosuppressive or myelosuppressive therapy with, e.g., monoclonal antibodies, methotrexate, cyclophosphamide, cyclosporine or azathioprine, or chronic use of corticosteroids.
15. Active malignancy or history of malignancy.
16. Received a live vaccine within 6 weeks prior to cladribine tablet administration or intends to receive a live vaccination during the trial. After the last dose of cladribine tablets, the subject should avoid live vaccine as long as the subject's white blood cell counts are not within normal limits.
17. Allergy or hypersensitivity to gadolinium and/or any other contraindication to perform an MRI.
18. Has any renal condition that would preclude the administration of gadolinium (e.g. acute or chronic severe renal insufficiency (GFR < 30 mL/min/1.73m2)

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Absolute and percent change of T cells, B cells, DC subset and NfL levels in blood. | 24 months
  The absolute and percent change from baseline will be presented for each time point for CD3+ T lymphocytes, CD19+ B lymphocytes, CD11c+ DC subsets, NfL levels in blood, with a two-sided 95% CI and p value. As these data are not expected to be normally distributed, the nonparametric Wilcoxon signed rank test will be used to compare each biomarker at baseline and during treatment. Spearman rank correlations will be used to examine the relationship between biomarkers and clinical/safety endpoints.

SECONDARY OUTCOMES:
Annualized Relapse Rate (ARR) | 12 months
  The ARR over the 12- and 24-month periods will be presented, accompanied by the respective 95% CIs. The proportion (and 95% CI) of participants experiencing a relapse over the 12 month and 24-month periods will also be presented.

OTHER OUTCOMES:
The Expanded Disability Status Scale : Neurological disability outcome | 24 months
  The Expanded Disability Status Scale (EDSS) will be utilized to measure the accumulation of neurological disability.
  The change in EDSS from baseline will be reported at month 12 and month 24. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
  EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems (FS):
  muscle weakness or difficulty moving limbs, ataxia, loss of balance, coordination or tremor, problems with speech, swallowing and nystagmus, numbness or loss of sensations, bowel and bladder function, problems with sight, problems with thinking and memory, other A functional system (FS) represents a network of neurons in the brain with responsibility for particular tasks. Each FS is scored on a scale of 0 (no disability) to 5 or 6 (more severe disability).
  EDSS steps 5.0 to 9.5 are defined by the impairment to walking.
Magnetic Resonance imaging (MRI) outcomes | 24 months
  The mean number of new or new/ enlarging T2 lesions, and the number of gadolinium (Gd)-enhancing lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Stuve, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - College Park Family Care Center Physicians Group, Overland Park, Kansas
  - UT Southwestern Medical center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartung HP, Graf J, Aktas O, Mares J, Barnett MH. Diagnosis of multiple sclerosis: revisions of the McDonald criteria 2017 - continuity and change. Curr Opin Neurol. 2019 Jun;32(3):327-337. doi: 10.1097/WCO.0000000000000699. PMID 30985371
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Shirani A, Stuve O. Natalizumab for Multiple Sclerosis: A Case in Point for the Impact of Translational Neuroimmunology. J Immunol. 2017 Feb 15;198(4):1381-1386. doi: 10.4049/jimmunol.1601358. PMID 28167648
- [Background] Shirani A, Stuve O. Natalizumab: Perspectives from the Bench to Bedside. Cold Spring Harb Perspect Med. 2018 Dec 3;8(12):a029066. doi: 10.1101/cshperspect.a029066. PMID 29500304
- [Background] Stuve O, Marra CM, Jerome KR, Cook L, Cravens PD, Cepok S, Frohman EM, Phillips JT, Arendt G, Hemmer B, Monson NL, Racke MK. Immune surveillance in multiple sclerosis patients treated with natalizumab. Ann Neurol. 2006 May;59(5):743-7. doi: 10.1002/ana.20858. PMID 16634029
- [Background] Stuve O, Marra CM, Bar-Or A, Niino M, Cravens PD, Cepok S, Frohman EM, Phillips JT, Arendt G, Jerome KR, Cook L, Grand'Maison F, Hemmer B, Monson NL, Racke MK. Altered CD4+/CD8+ T-cell ratios in cerebrospinal fluid of natalizumab-treated patients with multiple sclerosis. Arch Neurol. 2006 Oct;63(10):1383-7. doi: 10.1001/archneur.63.10.1383. PMID 17030653
- [Background] Stuve O, Cravens PD, Frohman EM, Phillips JT, Remington GM, von Geldern G, Cepok S, Singh MP, Tervaert JW, De Baets M, MacManus D, Miller DH, Radu EW, Cameron EM, Monson NL, Zhang S, Kim R, Hemmer B, Racke MK. Immunologic, clinical, and radiologic status 14 months after cessation of natalizumab therapy. Neurology. 2009 Feb 3;72(5):396-401. doi: 10.1212/01.wnl.0000327341.89587.76. Epub 2008 Nov 5. PMID 18987352
- [Background] del Pilar Martin M, Cravens PD, Winger R, Frohman EM, Racke MK, Eagar TN, Zamvil SS, Weber MS, Hemmer B, Karandikar NJ, Kleinschmidt-DeMasters BK, Stuve O. Decrease in the numbers of dendritic cells and CD4+ T cells in cerebral perivascular spaces due to natalizumab. Arch Neurol. 2008 Dec;65(12):1596-603. doi: 10.1001/archneur.65.12.noc80051. Epub 2008 Oct 13. PMID 18852339
- [Background] Yao K, Gagnon S, Akhyani N, Williams E, Fotheringham J, Frohman E, Stuve O, Monson N, Racke MK, Jacobson S. Reactivation of human herpesvirus-6 in natalizumab treated multiple sclerosis patients. PLoS One. 2008 Apr 30;3(4):e2028. doi: 10.1371/journal.pone.0002028. PMID 18446218
- [Background] Stuve O, Bennett JL. Pharmacological properties, toxicology and scientific rationale for the use of natalizumab (Tysabri) in inflammatory diseases. CNS Drug Rev. 2007 Spring;13(1):79-95. doi: 10.1111/j.1527-3458.2007.00003.x. PMID 17461891
- [Background] Cutter GR, Stuve O. Does risk stratification decrease the risk of natalizumab-associated PML? Where is the evidence? Mult Scler. 2014 Sep;20(10):1304-5. doi: 10.1177/1352458514531843. Epub 2014 May 8. PMID 24812045
- [Background] Berger JR, Fox RJ. Erratum to: Reassessing the risk of natalizumab-associated PML. J Neurovirol. 2016 Aug;22(4):536-537. doi: 10.1007/s13365-016-0431-x. No abstract available. PMID 27026534
- [Background] Berger JR, Fox RJ. Reassessing the risk of natalizumab-associated PML. J Neurovirol. 2016 Aug;22(4):533-5. doi: 10.1007/s13365-016-0427-6. Epub 2016 Feb 3. PMID 26843383
- [Background] Krumbholz M, Meinl I, Kumpfel T, Hohlfeld R, Meinl E. Natalizumab disproportionately increases circulating pre-B and B cells in multiple sclerosis. Neurology. 2008 Oct 21;71(17):1350-4. doi: 10.1212/01.wnl.0000327671.91357.96. PMID 18936427
- [Background] Kivisakk P, Healy BC, Viglietta V, Quintana FJ, Hootstein MA, Weiner HL, Khoury SJ. Natalizumab treatment is associated with peripheral sequestration of proinflammatory T cells. Neurology. 2009 Jun 2;72(22):1922-30. doi: 10.1212/WNL.0b013e3181a8266f. PMID 19487650
- [Background] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Background] Rudick RA, Stuart WH, Calabresi PA, Confavreux C, Galetta SL, Radue EW, Lublin FD, Weinstock-Guttman B, Wynn DR, Lynn F, Panzara MA, Sandrock AW; SENTINEL Investigators. Natalizumab plus interferon beta-1a for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):911-23. doi: 10.1056/NEJMoa044396. PMID 16510745
- [Background] Warnke C, Wiendl H, Hartung HP, Stuve O, Kieseier BC. Identification of targets and new developments in the treatment of multiple sclerosis--focus on cladribine. Drug Des Devel Ther. 2010 Jul 21;4:117-26. doi: 10.2147/dddt.s6627. PMID 20689698
- [Background] Carson DA, Kaye J, Seegmiller JE. Lymphospecific toxicity in adenosine deaminase deficiency and purine nucleoside phosphorylase deficiency: possible role of nucleoside kinase(s). Proc Natl Acad Sci U S A. 1977 Dec;74(12):5677-81. doi: 10.1073/pnas.74.12.5677. PMID 202960
- [Background] Carson DA, Wasson DB, Taetle R, Yu A. Specific toxicity of 2-chlorodeoxyadenosine toward resting and proliferating human lymphocytes. Blood. 1983 Oct;62(4):737-43. PMID 6136305
- [Background] Sipe JC. Cladribine tablets: a potential new short-course annual treatment for relapsing multiple sclerosis. Expert Rev Neurother. 2010 Mar;10(3):365-75. doi: 10.1586/ern.10.12. PMID 20187859
- [Background] Liliemark J. The clinical pharmacokinetics of cladribine. Clin Pharmacokinet. 1997 Feb;32(2):120-31. doi: 10.2165/00003088-199732020-00003. PMID 9068927
- [Background] Kawasaki H, Carrera CJ, Piro LD, Saven A, Kipps TJ, Carson DA. Relationship of deoxycytidine kinase and cytoplasmic 5'-nucleotidase to the chemotherapeutic efficacy of 2-chlorodeoxyadenosine. Blood. 1993 Feb 1;81(3):597-601. PMID 8094016
- [Background] Griffig J, Koob R, Blakley RL. Mechanisms of inhibition of DNA synthesis by 2-chlorodeoxyadenosine in human lymphoblastic cells. Cancer Res. 1989 Dec 15;49(24 Pt 1):6923-8. PMID 2573423
- [Background] Leist TP, Comi G, Cree BA, Coyle PK, Freedman MS, Hartung HP, Vermersch P, Casset-Semanaz F, Scaramozza M; oral cladribine for early MS (ORACLE MS) Study Group. Effect of oral cladribine on time to conversion to clinically definite multiple sclerosis in patients with a first demyelinating event (ORACLE MS): a phase 3 randomised trial. Lancet Neurol. 2014 Mar;13(3):257-67. doi: 10.1016/S1474-4422(14)70005-5. Epub 2014 Feb 4. PMID 24502830
- [Background] Giovannoni G, Comi G, Cook S, Rammohan K, Rieckmann P, Soelberg Sorensen P, Vermersch P, Chang P, Hamlett A, Musch B, Greenberg SJ; CLARITY Study Group. A placebo-controlled trial of oral cladribine for relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):416-26. doi: 10.1056/NEJMoa0902533. Epub 2010 Jan 20. PMID 20089960
- [Background] Giovannoni G, Soelberg Sorensen P, Cook S, Rammohan K, Rieckmann P, Comi G, Dangond F, Adeniji AK, Vermersch P. Safety and efficacy of cladribine tablets in patients with relapsing-remitting multiple sclerosis: Results from the randomized extension trial of the CLARITY study. Mult Scler. 2018 Oct;24(12):1594-1604. doi: 10.1177/1352458517727603. Epub 2017 Sep 5. PMID 28870107
- [Background] Leist TP, Vermersch P. The potential role for cladribine in the treatment of multiple sclerosis: clinical experience and development of an oral tablet formulation. Curr Med Res Opin. 2007 Nov;23(11):2667-76. doi: 10.1185/030079907x233142. PMID 17880754
- [Background] Kopadze T, Dehmel T, Hartung HP, Stuve O, Kieseier BC. Inhibition by mitoxantrone of in vitro migration of immunocompetent cells: a possible mechanism for therapeutic efficacy in the treatment of multiple sclerosis. Arch Neurol. 2006 Nov;63(11):1572-8. doi: 10.1001/archneur.63.11.1572. PMID 17101825
- [Background] Mitosek-Szewczyk K, Stelmasiak Z, Bartosik-Psujek H, Belniak E. Impact of cladribine on soluble adhesion molecules in multiple sclerosis. Acta Neurol Scand. 2010 Dec;122(6):409-13. doi: 10.1111/j.1600-0404.2010.01330.x. PMID 20175758
- [Background] Janiec K, Wajgt A, Kondera-Anasz Z. Effect of immunosuppressive cladribine treatment on serum leucocytes system in two-year clinical trial in patients with chronic progressive multiple sclerosis. Med Sci Monit. 2001 Jan-Feb;7(1):93-8. PMID 11208501
- [Background] De Stefano N, Giorgio A, Battaglini M, De Leucio A, Hicking C, Dangond F, Giovannoni G, Sormani MP. Reduced brain atrophy rates are associated with lower risk of disability progression in patients with relapsing multiple sclerosis treated with cladribine tablets. Mult Scler. 2018 Feb;24(2):222-226. doi: 10.1177/1352458517690269. Epub 2017 Jan 31. PMID 28140753
- [Background] Comi G, Cook SD, Giovannoni G, Rammohan K, Rieckmann P, Sorensen PS, Vermersch P, Hamlett AC, Viglietta V, Greenberg SJ. MRI outcomes with cladribine tablets for multiple sclerosis in the CLARITY study. J Neurol. 2013 Apr;260(4):1136-46. doi: 10.1007/s00415-012-6775-0. Epub 2012 Dec 21. PMID 23263473
- [Background] Comi G, Cook S, Rammohan K, Soelberg Sorensen P, Vermersch P, Adeniji AK, Dangond F, Giovannoni G. Long-term effects of cladribine tablets on MRI activity outcomes in patients with relapsing-remitting multiple sclerosis: the CLARITY Extension study. Ther Adv Neurol Disord. 2018 Jan 23;11:1756285617753365. doi: 10.1177/1756285617753365. eCollection 2018. PMID 29399054
- [Background] Freedman MS, Leist TP, Comi G, Cree BA, Coyle PK, Hartung HP, Vermersch P, Damian D, Dangond F. The efficacy of cladribine tablets in CIS patients retrospectively assigned the diagnosis of MS using modern criteria: Results from the ORACLE-MS study. Mult Scler J Exp Transl Clin. 2017 Oct 9;3(4):2055217317732802. doi: 10.1177/2055217317732802. eCollection 2017 Oct-Dec. PMID 29051829
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Meyer-Moock S, Feng YS, Maeurer M, Dippel FW, Kohlmann T. Systematic literature review and validity evaluation of the Expanded Disability Status Scale (EDSS) and the Multiple Sclerosis Functional Composite (MSFC) in patients with multiple sclerosis. BMC Neurol. 2014 Mar 25;14:58. doi: 10.1186/1471-2377-14-58. PMID 24666846